CLINICAL TRIAL: NCT06765200
Title: Effectiveness of a Digital Treatment for Adolescents with Chronic Pain
Acronym: DigiDOL-Ad
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Jordi Miró, Professor, University Rovira i Virgili
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PID2022-142071OB-I00
Record Dates: First submitted 2024-12-19; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; mhealth; adolescent; mobile application
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital treatment (Experimental): The treatment includes a smartphone-based psychosocial program designed to improve the quality of life of adolescents with chronic pain.
  Interventions: Behavioral: Self-administered psychosocial intervention delivered via smartphone.

INTERVENTIONS:
Behavioral: Self-administered psychosocial intervention delivered via smartphone. — The treatment includes a smartphone-based psychosocial program designed to improve the quality of life of adolescents with chronic pain.

SUMMARY:
Research has shown that the prevalence of chronic pain in adolescents is high and increasing. These young people report significant changes in both their physical and psychological functioning. Currently, psychosocial treatments enjoy strong empirical support and are crucial to maintaining and improving the quality of life of adolescents suffering from chronic pain. However, the availability of these evidence-based interventions is insufficient to meet the high demand, especially outside of large cities. The aim of this project is to develop a digital treatment that helps improve the quality of life of adolescents with chronic pain and complementary websites for their parents and teachers.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old,
* Having a non-oncology secondary chronic pain problem,
* Having internet access,
* A parent willing to participate in the study,
* Providing informed consent/assent.

Exclusion Criteria:

* Cognitive or language problems

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | baseline, 8 weeks, 3 months follow-up
  Refers to the severity of pain an individual experiences, measured on a scale (0-10)
Pain interference | baseline, 8 weeks, 3 months follow-up
  Refers to the extent to which pain affects an individual's daily life and functioning. Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Pain Interference will be used (0-32; 0=no interference, 32=intense interference).
Global perception of change after treatment | 8 weeks, 3 months follow-up
  refers to an individual's overall assessment of how their condition has improved or worsened following a treatment, measured on a scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Miró, Principal Investigator — University Rovira i Virgili
Locations (1):
- Universitat Rovira i Virgili, Tarragona, Spain

REFERENCES:
- [Derived] Miro J, Sampietro A, Monterde S, Ingelmo P, Wicksell RK, Nolla C, Alonso M, Lazaro JJ, Martinez E, Rubio P, Sanchez A, Sanchez V, Vazquez A, de la Vega R, Reinoso-Barbero F. Development, implementation and evaluation of a digital treatment for adolescents with chronic pain: a protocol for a multi-phase study. Front Digit Health. 2025 Jun 4;7:1555733. doi: 10.3389/fdgth.2025.1555733. eCollection 2025. PMID 40534825